CLINICAL TRIAL: NCT06744153
Title: Innovative Functional Space Maintainers Designed Using CAD/CAM Technology
Brief Title: Clinical Outcomes of Functional Space Maintainers Designed Using CAD/CAM Technology in Early Loss of the First Primary Molar
Acronym: KOS&MET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rasa Mladenovic (Other)
Responsible Party: Sponsor-Investigator, Rasa Mladenovic, Assistant professor, Pediatric dentist, University of Kragujevac
Organization: University of Kragujevac (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 01-14789/2022; Ethics Committee (Other: Faculty of Medical Sciences University of Kragujevac, Serbia)
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Dental Crowns; Orthodontics, Interceptive; Orthodontic Appliance
Keywords: functional space maintainers; CAD/CAM; 3D printing; Milling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D Print (Active Comparator): 3D Print (Metal) - Additive Method: In this group, the functional space maintainer was fabricated from a metal alloy (Co 69%, Cr 25%, W 9.5%, Mo 3.5%, Si 1%, Scheftner, Germany) using a 3D printer (MySint100 Dual Laser, Italy).
  Interventions: Procedure: Space Maintainer
- Milling (Active Comparator): Milling (Composite) - Subtractive Method: A dental milling machine (Wieland Zenotec Select Hybrid, Germany) was used to fabricate functional space maintainers from a polymer composite material (breCAM.HIPC, Bredent, Germany)
  Interventions: Procedure: Space Maintainer

INTERVENTIONS:
Procedure: Space Maintainer — Fabrication of KOS&MET functional space maintainer and its cementation.

SUMMARY:
As passive fixed space maintainers do not replace the lost tooth and therefore do not provide a chewing function, this study aims to evaluate the efficiency of an innovative solution for maintaining space after the premature extraction of first primary molars using functional space maintainers based on CAD/CAM technology.

DETAILED DESCRIPTION:
The innovative design of a functional space maintainer named KOS&MET (Key Orthodontic System and Materials Enhanced Therapy) was created using 3Shape Dental Designer (3Shape A/S, Copenhagen, Denmark). The functional maintainer features an intraoral window for monitoring the eruption of the successor tooth. In addition to its role in maintaining space, the maintainer is designed to restore bilateral chewing function. In addition to the loop encircling the second primary molar, the space maintainer includes a crown for the missing first primary molar. To achieve optimal anatomical details, we applied a mirror model of the molar from the contrary side.

Space maintainers were fabricated using CAD/CAM technology in two ways: 3D printing and milling.

1. 3D Print (Metal) - Additive Method: In this group, the functional space maintainer was fabricated from a metal alloy (Co 69%, Cr 25%, W 9.5%, Mo 3.5%, Si 1%, Scheftner, Germany) using a 3D printer (MySint100 Dual Laser, Italy).
2. Milling (Composite) - Subtractive Method: A dental milling machine (Wieland Zenotec Select Hybrid, Germany) was used to fabricate functional space maintainers from a polymer composite material (breCAM.HIPC, Bredent, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Indication for extraction or premature loss of the first primary molar in the upper or lower jaw.
* A prolonged time period from the loss of the primary tooth to the eruption of its successor (with bone tissue present above the successor tooth on the radiograph).
* A complete dental arch on the contrary side of the jaw.
* Intact or adequately restored vital second primary molars in the region indicated for the placement of a space maintainer.

Exclusion Criteria:

* Systemic disorders and uncooperative children.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical Evaluation - Fractures and decementing | 6 months
  The condition of the abutment teeth and surrounding soft tissues, as well as potential fractures or decementing of the space maintainer, were inspected at 1, 3, and 6 months.

SECONDARY OUTCOMES:
Bite Force (Newtone) | 1 Day
  Maximum Occlusal Bite Force in Newtones: Measured using a specially designed dynamometer (RABiter, Kragujevac, Serbia) directly on the space maintainer, with the contrary side of the jaw used as a control.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty od Medical Sciences University of Kragujevac, Kragujevac, Serbia

IPD SHARING:
Plan to Share IPD: No